CLINICAL TRIAL: NCT06722339
Title: Targeted Circuit-Based Transcranial Focused Ultrasound Intervention for Obsessive-Compulsive Disorder
Brief Title: Targeted Circuit-Based Transcranial Focused Ultrasound Intervention for Obsessive-Compulsive Disorder TUS-OCD
Acronym: TUS-OCD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Elsa Fouragnan, Associate Professor, University of Plymouth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 2024-4821-6128; MR/T023007/1 (Other Grant/Funding Number: UKRI MRC)
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: focused ultrasound; TUS; neuromodulation; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Within subject, randomized, double-blind, sham-controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TUS sham (Other): double-blind, sham-controlled, crossover study in N=30 individuals with OCD
  Interventions: Device: low intensity transcranial focused ultrasound stimulation (TUS)
- TUS Active (Other): double-blind, sham-controlled, crossover study in N=30 individuals with OCD
  Interventions: Device: low intensity transcranial focused ultrasound stimulation (TUS)

INTERVENTIONS:
Device: low intensity transcranial focused ultrasound stimulation (TUS) — Low-intensity transcranial focused ultrasound (TUS) provides an energy source with millimeter resolution that can be focused anywhere in the brain safely and effectively for non-invasive and transient neuromodulation. TUS is an important advance and of great significance for brain-mapping efforts, diagnostics, and therapies in neuroscience and particularly promising for addiction therapy as it provides unprecedented non-surgical access to the brain regardless of depth.
  Low intensities of focused ultrasound (TUS) are used so that tissue damage does not occur, but neural activity can be modulated by mechanical effects.
  Other Names: low intensity focused ultrasound (LIFU)

SUMMARY:
This study explores the potential of transcranial ultrasound stimulation (TUS) as an innovative therapeutic approach for individuals with obsessive-compulsive disorder (OCD). By targeting specific brain regions associated with compulsive behaviors and anxiety, the researchers aim to assess the safety and efficacy of TUS in reducing symptoms and enhancing cognitive flexibility.

DETAILED DESCRIPTION:
Obsessive Compulsive Disorder (OCD) is a common and highly debilitating disorder with the manifestation of obsessions/compulsions and is associated with a significant impairment in social functioning and quality of life. Estimates show that the effects of OCD create an economic burden of £5 billion/year in the UK alone (Kochar et al. 2023). Novel interventions with greater efficacy in addressing the symptoms of OCD in patients, aiming to surpass the current standards of effectiveness and comprehensiveness in treatment outcomes are needed. Low-intensity transcranial focused ultrasound stimulation (TUS) is a promising emerging non-invasive brain stimulation technique which can neuromodulate any brain region with high spatial resolution.

The neural underpinning of OCD is thought to involve many prefrontal regions including the anterior cingulate cortex (ACC) but also deeper brain regions like the striatum (habit formation: Ahmari et al. 2017, Denys et al. 2013), the thalamus (Subirà et al. 2016) and the amygdala (overactivity: Fullana et al. 2020, Milad et al. 2013). TUS can focally induce changes in neuronal activity in both cortical and subcortical brain regions with incredibly high spatial resolution (Darmani et al. 2022). The current study will focus on targeting multiple regions playing a significant role in regulating various cognitive and repeated actions in OCD. We will assess safety and efficiency of TUS to different parts of the brain in alleviating OCD symptoms.

ELIGIBILITY:
Inclusion Criteria will be:

* Male or female, aged 21-55 years, and fluent English speaking.
* Participants score ≥ 17 on the Obsessive-Compulsive Inventory-Revised (OCI-R).
* Participant is willing and able to give informed consent for participation in the trial.
* Participant is willing to comply with all trial requirements and committed to participating in all six testing sessions.

Exclusion Criteria will be:

The participant may not enter the trial if ANY of the following apply.

History:

* serious head trauma or brain surgery
* (first-degree relatives with) epilepsy, convulsion, or seizure
* diagnosis of a neurological or psychiatric disorder (other than OCD)
* adverse reactions to non-invasive brain stimulation
* participation in another short-term non-invasive brain stimulation study in the past 3 days
* participation in another long-term non-invasive brain stimulation study in the past 28 days
* recent head trauma that was diagnosed as a concussion or associated with loss of consciousness

Current:

* pregnancy or planning a pregnancy during the course of the trial
* use of psychoactive drugs or any drugs listed in the Neurostimulation Safety Report
* heart pacemaker, mechanical heart valve, mechanical implant such as an aneurysm clip, hip replacement
* metal in the head or body
* claustrophobia
* extreme mood fluctuations
* predisposition to fainting spells (syncope)
* medication that will interfere with the study or constitutes an increased risk of adverse effects (e.g., affects brain excitability)
* hearing problems or ringing in the ears
* skin diseases or sensitivity at intended TUS stimulation site
* Any significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Last 24 hours:

* more than four alcoholic units
* recreational psychoactive drugs
* antibiotics

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-09-19 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Immediately after TUS session; one day and one week after TUS. Same for sham, to compare the TUS active and sham.
  number of adverse events

SECONDARY OUTCOMES:
reduction in OCD symptoms | immediately prior to TUS sessions, within 1 hour post TUS and every day that follow TUS for 7 days
  numerical OCD symptoms rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Elsa F Fouragnan, Ph.D., Principal Investigator — University of Plymouth
Locations (1):
- Health, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymous behavioral data upon publication
Supporting Information: SAP, Analytic Code
Time Frame: data will be available after analysis of primary and secondary outcomes are completed
Access Criteria: anyone with access to the link to the data (OSF)
URL: http://www.plymouth.ac.uk/students-and-family/governance/general-data-protection-regulation-gdpr

REFERENCES:
- See also: safety report for TUS use from expert consortium — https://arxiv.org/abs/2311.05359